CLINICAL TRIAL: NCT05260359
Title: Evaluation Bemotrizinol in Human Repeated Insult Patch Test (HRIPT) and Cumulative Irritation Test
Brief Title: Dermal Irritation, Sensitization and Cumulative Irritation Potential of 6% Bemotrizinol
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: DSM RIPT 2020
Record Dates: First submitted 2022-02-11; First posted 2022-03-02 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Sunburn
Keywords: cumulative irritation; irritation; sensitization; Bemotrizinol; Sunscreen
MeSH Terms: conditions — Sunburn | interventions — bis-ethylhexyloxyphenol methoxyphenyl triazine; Petrolatum; Sunscreening Agents; Ethanol; Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: A 21-Day controlled study to evaluate the skin Irritation and sensitization potential of 6% Bemotrizinol (BEMT) in topical products with vehicle controls after repeated patch applications to healthy human participants by following conventional Repeated Insult (HRIPT) and Cumulative Irritation (CIT) methodologies.
Who Masked: Participant
Masking Description: Subjects will be blinded to the name of the investigational products
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 6% BEMT HRIPT (Active Comparator): During the challenge phase of the HRIPT portion of the study, there will be 6 patches (2 product patches, 2 vehicle controls. 1 saline control and 1 empty patch), leaving out the positive control.
  Interventions: Drug: 6% Bemotrizinol (BEMT) in a basic sunscreen oil formulation; Drug: 6% Bemotrizinol (BEMT) dispersion in petrolatum; Other: Sunscreen oil vehicle with 10% ethanol as penetration enhancer without BEMT; Other: Petrolatum vehicle; Other: 0.9% Saline; Other: Undosed patch
- 6% BEMT Cumulative Irritation Study (Active Comparator): During the Cumulative Irritation portion of the study there will be 7 patches (2 product patches, 2 vehicle controls, 1 positive control, 1 low-irritancy control, and 1 empty patch). The low-irritancy control patch will be a saline patch. The positive control will be a SLS patch. The negative control will be an undosed patch.
  Interventions: Drug: 6% Bemotrizinol (BEMT) in a basic sunscreen oil formulation; Drug: 6% Bemotrizinol (BEMT) dispersion in petrolatum; Other: Sunscreen oil vehicle with 10% ethanol as penetration enhancer without BEMT; Other: Petrolatum vehicle; Other: 0.9% Saline; Other: Sodium Lauryl Sulfate 0.1% (SLS); Other: Undosed patch

INTERVENTIONS:
Drug: 6% Bemotrizinol (BEMT) in a basic sunscreen oil formulation — SU E 101413 85
  Other Names: PARSOL® SHIELD
Drug: 6% Bemotrizinol (BEMT) dispersion in petrolatum — SU-E-101413-82
  Other Names: PARSOL® SHIELD
Other: Sunscreen oil vehicle with 10% ethanol as penetration enhancer without BEMT — SU E 101413 91
  Other Names: Sunscreen oil Vehicle
Other: Petrolatum vehicle — SU-E-101413-83
  Other Names: Vehicle
Other: 0.9% Saline — low irritancy control
  Other Names: Saline
Other: Sodium Lauryl Sulfate 0.1% (SLS) — positive control
  Other Names: control
  Arms: 6% BEMT Cumulative Irritation Study
Other: Undosed patch — negative control
  Other Names: control

SUMMARY:
The purpose of this clinical trial is to evaluate the dermal safety of Bemotrizinol (6%).

DETAILED DESCRIPTION:
The first objective of this study is to determine if 6% Bemotrizinol (BEMT) either in a basic sunscreen oil formulation (SU E 101413 85) or as dispersion in petrolatum (SU-E-101413-82) elicit dermal irritation and/or induce sensitization following repeated patch application.

The second objective of this study is to determine the cumulative irritation potential of 6% BEMT either in a basic sunscreen oil formulation (SU E 101413 85) or as dispersion in petrolatum (SU-E-101413-82) topically applied to the skin of human subjects over a 21-day period via a Human Repeat Insult Patch Test (HRIPT).

HRIPT: This part of the study will consist of an Induction Phase, a Challenge Phase, and, at the discretion of the Principal Investigator, a Re-Challenge Phase. During the Induction Phase, the test material will be applied to the same location on the back of each subject three times per week for a total of nine applications with 24 to 48 hour rest periods. Test sites will be examined for dermal irritation at each visit prior to reapplication of the test material. Approximately 14 days after the final visit of the Induction Phase, subjects will return to the laboratory for the Challenge Phase. The test material will be applied to a naïve site on the back under an appropriate patch and will be removed by clinical staff approximately 24 hours later. Test sites will be examined for signs of dermal irritation or sensitization. A subject may be required to return to the laboratory for a Re-Challenge Test, if reactions indicative of sensitization are observed during the Challenge Phase. During the Re-Challenge Phase, the test material will be applied to a naïve site under the same conditions of the Challenge Phase, and the subject will be examined for dermal reactions.

Cumulative Irritation Study: A subset of individuals selected for the HRIPT study will also participate in the Cumulative Irritation Study. Subjects who meet inclusion and exclusion criteria will be enrolled. Subjects will be consented and screened to determine eligibility and qualified subjects will be enrolled. Subjects will participate in a 21-day cumulative irritation patch study on the back. Test products and vehicle patches, along with a high irritancy, a low irritancy and empty patch controls, will be tested during the study.

At the Day 1 Visit, the upper back of each subject (between the scapulae to either side of the spinal midline) will be wiped with 70% isopropyl alcohol and allowed to dry. The empty patch, low irritancy 0.9% Saline control and the high irritancy Sodium Lauryl Sulfate 0.1% (SLS) control will be used as negative and positive controls, respectively. Controls and test products will be applied to the back daily, for approximately 21 days. Patches will remain in place for a period of approximately 24 hours. Test sites will be graded following each patch removal.

The vehicle controls (SU E 101413 91 and SU-E-101413-83), 0.9% saline and empty patches as negative control will be used for the HRIPT and Cumulative Irritation portion of the study. The 0.1% Sodium Laurel Sulfate (SLS) will be only used for the Cumulative Irritation portion of the study.

Approximately 0.2 g of the investigational products and the vehicle control will each be applied to the fabric portion of separate patches.

During the Cumulative Irritation portion of the study, there will be 7 patches (2 product patches, 2 vehicle controls, 1 positive control, 1 low-irritancy control, and 1 empty patch). The low-irritancy control patch will be a saline patch. The positive control will be a SLS patch. The negative control will be an undosed patch.

During the challenge phase of the HRIPT portion of the study, there will be 6 patches (2 product patches, 2 vehicle controls. 1 saline control and 1 empty patch), leaving out the positive control.

The patches to be used for this clinical trial will be occlusive strips (manufactured by Strukmyer LLC, Mesquite, TX or equivalent), consisting of a breathable tape with non- breathable adhesive and center portion of 1.9 cm x 1.9 cm fabric.

Dermal scores will be reported for each site.

Safety of the investigational products will be monitored by evaluating adverse event reporting.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female between 18 and 75 years of age;
2. Subject does not exhibit any skin diseases or abnormalities which might be confused with a skin reaction from the test material;
3. Subject agrees to avoid excessive sun exposure of the test sites and to refrain from visits to tanning salons during the course of this study;
4. Subject agrees to refrain from getting patches wet, scrubbing or washing the test area with soap, and applying powders, lotions or personal care products to the area during the course of the study;
5. Subject agrees not to introduce any new cosmetic or toiletry products during the study;
6. Subject is dependable and able to follow directions as outlined in the protocol;
7. Subject is willing to participate in all study evaluations;
8. Subject is in generally good health and has a current Panelist Profile Form and Medical History Form on file at CRL;
9. Subject has completed a HIPAA Authorization Form in conformance with 45 code of federal regulation (CFR) Parts 160 and 164;
10. Subject understands and is willing to sign an Informed Consent Form in conformance with 21 CFR Part 50: "Protection of Human Subjects."

Exclusion Criteria:

1. Female subject is pregnant, nursing, planning a pregnancy, or not using adequate birth control;
2. Subject has a known allergy to any of the formulation ingredients; Ingredients INCI names: BIS-ETHYLHEXYLOXYPHENOL METHOXYPHENYL TRIAZINE; ALCOHOL; C12-15 ALKYL BENZOATE; CAPRYLIC/CAPRIC TRIGLYCERIDE; DICAPRYLYL CARBONATE; ISOPROPYL MYRISTATE; PETROLATUM; PHENETHYL BENZOATE;
3. Subject has received treatment with sympathomimetics, antihistamines, vasoconstrictors, non-steroidal anti-inflammatory agents, and/or systemic or topical corticosteroids within one week prior to initiation of the study;
4. Subject has a history of acute or chronic dermatologic (including active eczema or psoriasis on the test sites), medical, and/or physical conditions which would preclude application of the test material and/or could influence the outcome of the study;
5. Subject is under treatment for a skin and/or systemic bacterial infection;
6. Subject has scheduled, or is planning to undergo, any medical or surgical procedures during the 7 week course of the study
7. Subject exhibits birthmarks, moles, vitiligo, keloids, or any dermal markings on the back that might interfere with grading;
8. Subject has a known communicable disease (e.g., HIV, sexually transmitted diseases, Hepatitis B, Hepatitis C, etc.);
9. Subject is an insulin-dependent diabetic;
10. Subject has a history of skin cancer or is currently undergoing treatment for active cancer of any type;
11. Subject reports a history of allergies to tape adhesives;
12. Subject is currently taking certain medications which, in the opinion of the Principal Investigator, may interfere with the study;
13. Subject has known allergies to skin treatment products or cosmetics, toiletries, and/or topical drugs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2022-04-08 (Actual)

PRIMARY OUTCOMES:
Determine the dermal irritation (erythema) potential of 6% BEMT over 21 days | 21 days
  Dermal irritation and/or sensitization rated based on following scoring system:
  0 - No evidence of irritation
  1. - Minimal erythema, barely perceptible
  2. - Definite erythema, readily visible; minimal edema or minimal papular response
  3. - Erythema and papules
  4. - Definite edema
  5. - Erythema, edema, and papules
  6. - Vesicular eruption
  7. - Strong reaction spreading beyond test site
Determine the dermal sensitization potential of 6% BEMT after 24 hours | 24 hours
  After a 14 day rest period, a challenge test will be given to look at signals of a sensitization response measured by using the following scoring system:
  0 - No evidence of irritation
  1. - Minimal erythema, barely perceptible
  2. - Definite erythema, readily visible; minimal edema or minimal papular response
  3. - Erythema and papules
  4. - Definite edema
  5. - Erythema, edema, and papules
  6. - Vesicular eruption
  7. - Strong reaction spreading beyond test site
Determine the dermal sensitization potential of 6% BEMT after 48 hours | 48 hours
  After a 14 day rest period, a challenge test will be given to look at signals of a sensitization response measured by using the following scoring system:
  0 - No evidence of irritation
  1. - Minimal erythema, barely perceptible
  2. - Definite erythema, readily visible; minimal edema or minimal papular response
  3. - Erythema and papules
  4. - Definite edema
  5. - Erythema, edema, and papules
  6. - Vesicular eruption
  7. - Strong reaction spreading beyond test site
Determine the dermal sensitization potential of 6% BEMT after 72 hours | 72 hours
  After a 14 day rest period, a challenge test will be given to look at signals of a sensitization response measured by using the following scoring system:
  0 - No evidence of irritation
  1. - Minimal erythema, barely perceptible
  2. - Definite erythema, readily visible; minimal edema or minimal papular response
  3. - Erythema and papules
  4. - Definite edema
  5. - Erythema, edema, and papules
  6. - Vesicular eruption
  7. - Strong reaction spreading beyond test site
Determine the dermal sensitization potential of 6% BEMT after 96 hours | 96 hours
  After a 14 day rest period, a challenge test will be given to look at signals of a sensitization response measured by using the following scoring system:
  0 - No evidence of irritation
  1. - Minimal erythema, barely perceptible
  2. - Definite erythema, readily visible; minimal edema or minimal papular response
  3. - Erythema and papules
  4. - Definite edema
  5. - Erythema, edema, and papules
  6. - Vesicular eruption
  7. - Strong reaction spreading beyond test site
Determine the cumulative irritation potential of 6% BEMT over 21 days | 21 days
  The cumulative irritation potential of 6% bemotrizinol (BEMT) will be assessed for each subject via a visual assessment of the test products and controls during a 21-day application period. Cumulative irritation potential will be assessed using the following scoring system:
  0 - No evidence of irritation
  1. - Minimal erythema, barely perceptible
  2. - Definite erythema, readily visible; minimal edema or minimal papular response
  3. - Erythema and papules
  4. - Definite edema
  5. - Erythema, edema, and papules
  6. - Vesicular eruption
  7. - Strong reaction spreading beyond test site

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Poweski, Principal Investigator — Eurofins CRL Inc.
Locations (1):
- Eurofins | CRL, Inc., Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McNamee PM, Api AM, Basketter DA, Frank Gerberick G, Gilpin DA, Hall BM, Jowsey I, Robinson MK. A review of critical factors in the conduct and interpretation of the human repeat insult patch test. Regul Toxicol Pharmacol. 2008 Oct;52(1):24-34. doi: 10.1016/j.yrtph.2007.10.019. Epub 2007 Dec 4. PMID 18639964
- [Background] Api AM, Vey M. Implementation of the dermal sensitization Quantitative Risk Assessment (QRA) for fragrance ingredients. Regul Toxicol Pharmacol. 2008 Oct;52(1):53-61. doi: 10.1016/j.yrtph.2008.05.011. Epub 2008 May 27. PMID 18635300
- See also: Department of Health and Human Services, Food and Drug Administration, Center for Drug Evaluation and Research. Guidance for Industry: Nonprescription Sunscreen Drug Products - Safety and Effectiveness Data. — https://www.fda.gov/media/94513/download
- See also: U.S. Department of Health and Human Services. Assessing the Irritation and Sensitization Potential of Transdermal and Topical Delivery Systems for ANDAs: Guidance for Industry. 2018. — https://www.fda.gov/media/117569/download